CLINICAL TRIAL: NCT04238832
Title: Impact of Non-Cigarette Tobacco Product Formulation on Reinforcement Value and Use in Current Smokers
Brief Title: Salt-Based E-cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Tracy Smith, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00093724
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the staff nor the participants will be told whether the e-liquid is free base or salt based.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Base Nicotine (Active Comparator): Participants assigned to this group will try both a free base nicotine and a salt base nicotine, and then take home an e-cigarette and free base nicotine e-liquid to sample for one week.
  Interventions: Other: Free Base Nicotine
- Salt Base Nicotine (Active Comparator): Participants assigned to this group will try both a free base nicotine and a salt base nicotine, and then take home an e-cigarette and salt base nicotine e-liquid to sample for one week.
  Interventions: Other: Salt Base Nicotine

INTERVENTIONS:
Other: Salt Base Nicotine — Participants will try both free base and salt base nicotine e-liquid and then take home salt base nicotine
  Arms: Salt Base Nicotine
Other: Free Base Nicotine — Participants will try both free base and salt base nicotine e-liquid and then take home free base nicotine
  Arms: Free Base Nicotine

SUMMARY:
Electronic nicotine delivery systems (ENDS) vary on a wide range of characteristics, which may impact the reinforcement value of the products compared to more harmful combustible products. A new type of low-powered ENDS device has surged in popularity-the pod system. Pods use nicotine salt e-liquids, rather than free-base nicotine solutions that have been used in other ENDS device types. Manufacturers claim that these formulations reduce the harshness of nicotine delivery, while still delivering sufficiently high levels of nicotine. However, the role of nicotine salts in the popularity and use of pod systems remains unclear because no studies have directly manipulated and examined the role of nicotine formulation (salt vs. free base) in reinforcement value and use. The primary purpose of the proposed study is to assess the impact of nicotine formulation (nicotine salt vs. free-base) in reinforcement value and tobacco use. Current smokers (n=30) will complete a one-week baseline period where they smoke as normal before attending an in-person lab visit during which they will sample a traditional cigarette and two ENDS products (nicotine salt ENDS, free base ENDS). All aspects of the device will be held constant other than the nicotine formulation (including nicotine concentration, flavor options, device brand). Participants will answer questionnaires about each product they sample and then complete a preference assessment in which they choose between the products they sampled and their own cigarette. Finally, participants will be assigned to take one of the products they sampled home to use ad libitum (1-week sampling). During the at-home baseline and sampling weeks, participants will complete electronic daily diaries cataloging their tobacco use. Biomarkers (i.e., expired carbon monoxide, cotinine) will corroborate self-reported indices of use.

ELIGIBILITY:
Inclusion Criteria:

* daily cigarette smoker
* interested in using non-cigarette tobacco product
* have a smartphone that can receive text messages and has access to the internet or have an e-mail account they check daily (necessary for daily diary completion).

Exclusion Criteria:

* additional tobacco use criteria
* additional medical criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Most preferred product | Lab Visit 2, occurring approximately one week after the initial screening/baseline visit
  Participants complete a preference assessment in which they choose between the salt liquid, free base liquid, or a traditional cigarette in a series of trials. The outcome of this assessment is the product chosen most often by each participant.

SECONDARY OUTCOMES:
Cigarettes per day | Week 2 of study
  The average number of cigarettes smoked per day during the one week sampling period

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided